CLINICAL TRIAL: NCT00289822
Title: Cell Therapy for Coronary Heart Disease: Infusion of Autologous Ex Vivo Cultivated Endothelial Progenitor Cells (EPCs)" and Autologous Bone Marrow Progenitor Cells in Crossover Design for Improvement of Vascularization and Cardiac Function
Brief Title: Cell Therapy for Coronary Heart Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 158/02
Record Dates: First submitted 2006-02-08; First posted 2006-02-10 (Estimated); Last update posted 2006-11-30 (Estimated); Status verified 2006-02

CONDITIONS: Coronary Artery Disease
Keywords: chronic heart failure; myocardial infarction
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Infarction

INTERVENTIONS:
Drug: intracoronary infusion of progenitor cells

SUMMARY:
Impaired contractile function after a heart attack and due to coronary heart disease is a major cause of "heart failure" limiting quality of life and prognosis, which cannot be prevented even with optimal standard therapy.

The aim of the current trial is to investigate whether infusion of progenitor cells into the coronary artery supplying the most dyskinetic left ventricular area may improve left ventricular contractile function, compared to no cell infusion in the control group, in patients with old (>= 3 months) myocardial infarction.

DETAILED DESCRIPTION:
* The study is an open-label, controlled, randomized single-center trial.
* Patients post myocardial infarction (>= 3 months) with a patent infarct-related artery are included.
* Bone marrow-derived progenitor cells are aspirated under local anaesthesia, and after cell processing, are infused into the patent infarct-related artery during stop flow within the same day. Blood-derived progenitor cells are isolated out of 250ml peripheral venous blood, and after cell processing and 3 days culture, are infused into the patent infarct-related artery during stop flow. In addition, left ventricular angiography is performed. In the control group coronary angiography and left ventricular angiography without any intracoronary infusion are performed.
* After 3 months, left ventricular angiography is repeated, and patients of the control group cross-over to active treatment with progenitor cells, whereas patients initially treated with progenitor cells cross-over to the alternate cell type.
* The primary endpoint is the change in quantitative global left ventricular ejection fraction in LV angiography between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 80
* Patients post-myocardial infarction (> 3 months old) or with diffuse ischemic CHD
* Signed informed consent

Exclusion Criteria:

- Existing neoplastic disease or signs of tumor recurrence within the last 5 years

* Active infection
* Active internal bleeding
* Stroke within the past 2 years
* Surgery or trauma within the past two months
* Uncontrolled hypertension over 160/100
* Arteriovenous malformations or aneurysms
* HIV infection
* Signs of significant kidney or liver failure (creatinine > 2.0 mg/dL, GOT > 2 x upper standard value)
* Thrombopenia (< 100,000)
* Anemia (hemoglobin < 8.5 g/dL)
* Mental retardation
* Participation in another clinical study
* Women of childbearing age
* Chronic inflammatory disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75
Dates: Start 2002-01; Study Completion 2005-01

PRIMARY OUTCOMES:
Change in global left ventricular function (measured by quantitative left ventricular angiography)

SECONDARY OUTCOMES:
Quantitative parameters of regional left ventricular function of the target area
changes in left ventricular volumes
functional status as assessed by NYHA classification
event-free survival after 4 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Andreas M Zeiher, MD, Principal Investigator — J. W. Goethe University Hospitals; Volker Schaechinger, MD, Study Director — J. W. Goethe University Hospitals
Locations (1):
- J. W. Goethe University Hospitals, Frankfurt, Germany

REFERENCES:
- [Result] Assmus B, Honold J, Schachinger V, Britten MB, Fischer-Rasokat U, Lehmann R, Teupe C, Pistorius K, Martin H, Abolmaali ND, Tonn T, Dimmeler S, Zeiher AM. Transcoronary transplantation of progenitor cells after myocardial infarction. N Engl J Med. 2006 Sep 21;355(12):1222-32. doi: 10.1056/NEJMoa051779. PMID 16990385
- [Derived] De Rosa S, Seeger FH, Honold J, Fischer-Rasokat U, Lehmann R, Fichtlscherer S, Schachinger V, Dimmeler S, Zeiher AM, Assmus B. Procedural safety and predictors of acute outcome of intracoronary administration of progenitor cells in 775 consecutive procedures performed for acute myocardial infarction or chronic heart failure. Circ Cardiovasc Interv. 2013 Feb;6(1):44-51. doi: 10.1161/CIRCINTERVENTIONS.112.971705. Epub 2013 Jan 29. PMID 23362308
- [Derived] Leistner DM, Seeger FH, Fischer A, Roxe T, Klotsche J, Iekushi K, Seeger T, Assmus B, Honold J, Karakas M, Badenhoop K, Frantz S, Dimmeler S, Zeiher AM. Elevated levels of the mediator of catabolic bone remodeling RANKL in the bone marrow environment link chronic heart failure with osteoporosis. Circ Heart Fail. 2012 Nov;5(6):769-77. doi: 10.1161/CIRCHEARTFAILURE.111.966093. Epub 2012 Aug 30. PMID 22936827